CLINICAL TRIAL: NCT04553666
Title: Reducing Frailty for Older Cancer Survivors Using Supplements (ReFOCUS): A Phase 2 Randomized Controlled Trial of Epigallocatechin-3-Gallate (EGCG) on Frailty and Inflammation in Older Survivors of Cancer
Brief Title: Reducing Frailty for Older Cancer Survivors Using Supplements
Acronym: ReFOCUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Nikesha Gilmore, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS20081
Record Dates: First submitted 2020-09-04; First posted 2020-09-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Frailty; Inflammation
MeSH Terms: conditions — Frailty; Inflammation | interventions — epigallocatechin gallate; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Patients in the intervention Arm will receive 800 mg Epigallocatechin gallate (EGCG) + 250mg Ascorbic Acid
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Four 200mg EGCG pills and one 250mg Vitamin C pill taken one time each day
  Interventions: Drug: Epigallocatechin-3-Gallate (EGCG) plus Ascorbic Acid (Vitamin C)
- Usual Care Group (No Intervention): No study pills

INTERVENTIONS:
Drug: Epigallocatechin-3-Gallate (EGCG) plus Ascorbic Acid (Vitamin C) — 800mg Epigallocatechin-3-Gallate (EGCG) plus 250mg Ascorbic Acid (Vitamin C) taken one time a day for twelve weeks
  Other Names: EGCG plus Vitamin C
  Arms: Intervention Group

SUMMARY:
The purpose of the study is to examine the feasibility and safety of twelve weeks oral supplementation of Epigallocatechin-3-gallate (EGCG) in older survivors of cancer

ELIGIBILITY:
Inclusion Criteria:

1. Be age 65 or over.
2. Be diagnosed with stage I-III Cancer.
3. Have completed curative intent treatment ≤10 years prior to screening. (Patients on endocrine therapies are allowed to enroll.)
4. Have a Fried's Frailty Score (FFS) of ≥ 2.
5. Able to provide informed consent, or have consent given by patient-designated health care proxy per institutional policies and University of Rochester Cancer Control guidelines.

Exclusion Criteria: Study subjects must not:

1. Have chemotherapy planned for the during of the study.
2. Have abnormal liver function tests (ALT, AST and bilirubin ≥3 times institutional upper limit of normal) per most recent available lab test (within 3 months of screening).
3. Have uncontrolled or unmanaged liver disease.
4. Consume more than 6 cups of green tea per day.
5. Have known allergies to caffeine.
6. Be diagnosed with a major psychiatric illness requiring hospitalization within the last year.
7. Be diagnosed with dementia.
8. Cannot provide informed consent due to lack of decision making capacity (as determined by the patient's oncologist) and has no patient-designated health care proxy per institutional policies and University of Rochester Cancer Control URCC guidelines.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from clinical sites within Wilmot Cancer Institute between April 2021 and March 2023. Eligible patients were aged 65 or older, diagnosed with Stage I-III solid cancer, completed curative intent treatment 10 years or less before being screened, and had a Fried's Frailty Score (FFS ≥ 2); assessed by measuring grip strength, weight loss, physical activity, fatigue, and a 4-meter walk test. The first participant was consented on April 28, 2021, and randomized on May 6, 2021.
Pre-assignment Details: Sixty four (64) potentially eligible participants were approached and 24 participants were consented. Of the 24 consented subjects: 5 screen failed (participant was consented but didn't fully meet eligibility criteria e.g. meet frailty cut off or liver toxicity screen); 4 screen withdrew (participant was consented but withdrew from the study before the baseline visit for randomization), and 1 was lost to follow up. Fourteen (14) participants were randomized to the treatment groups.
Groups:
- Usual Care Group: No study pills. Followed Usual Care procedures for a survivor of cancer according to oncology care teams' directions.
Period: Overall Study
Arm/Group | Intervention Group | Usual Care Group
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 14 subjects whose baseline measurements were received.
Groups:
- Usual Care Group: No study pills. Followed Usual Care procedures for an older survivor of cancer according to oncology care teams' directions.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Usual Care Group | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Customized [Mean (Full Range); unit: years]
  Age, Years: Mean | 76.6 [65 to 90] | 72.6 [66 to 80] | 74.5 [65 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  Some College | 1 | 2 | 3
  College and Above | 6 | 5 | 11
Marital Status [Count of Participants; unit: Participants]
  Married | 4 | 5 | 9
  Unmarried | 3 | 2 | 5
Employment Status [Count of Participants; unit: Participants]
  Retired | 6 | 6 | 12
  Employed | 1 | 1 | 2
Cancer Stage [Count of Participants; unit: Participants] — Cancer stage was reviewed from the patient's medical records and confirmed with their provider to ensure eligibility.
  Stage 0: abnormal cells are present and have not spread to nearby tissue. Stage 1: the cancer is small and contained within the organ it started in. Stage 2: the cancer has grown and possibly spread to nearby lymph nodes. Stage 3: the cancer has grown more and has spread to surrounding tissues including nearby lymph nodes.
  Stage 4: the cancer had spread to distant parts of the body.
  Participants
    Stage I | 4 | 3 | 7
    Stage II | 2 | 3 | 5
    Stage III | 1 | 1 | 2
Cancer Type [Count of Participants; unit: Participants]
  Colon/Rectal/Anal | 4 | 3 | 7
  Breast | 3 | 3 | 6
  Prostate | 0 | 1 | 1
Cancer Treatment [Count of Participants; unit: Participants]
  Surgery Alone | 2 | 3 | 5
  Surgery with Chemotherapy | 2 | 3 | 5
  Surgery with Radiation | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility: Rates of Consent
Description: Recruitment feasibility will be determined by the proportion of participants approached compared to those consented onto the study.
Time Frame: Baseline
Population: Since this outcome measure looks at the number of participants approached versus consented, the number of participants analyzed was the 64 approached instead of the 14 that were randomized.
Measure: Number; unit: proportion of participants
Groups:
- Proportion of Participants Consented: Proportion of participants approached compared to those consented onto the study
Arm/Group | Proportion of Participants Consented
Number analyzed (Participants) | 64
proportion of participants | 0.375

2. Primary Outcome: Recruitment Feasibility: Rates of Randomization
Description: Recruitment feasibility will be determined by the proportion of participants consented compared to those randomized into one of the study arms.
Time Frame: Baseline
Population: Since this outcome measure looks at the number of participants consented versus randomized, the number of participants analyzed was the 24 consented instead of the 14 that were randomized.
Measure: Number; unit: proportion of participants
Groups:
- Proportion of Participants Randomized: Proportion of participants consented compared to those randomized onto the study
Arm/Group | Proportion of Participants Randomized
Number analyzed (Participants) | 24
proportion of participants | 0.583

3. Primary Outcome: The Proportion of Participants That Completed the Study
Description: To determine adherence of a two arm randomized clinical trial of EGCG supplementation in older survivors of cancer by determining how many participants completed the study.The number of participants randomized compared to the number of participants that returned for the post intervention visit.
Time Frame: 12 week
Measure: Number; unit: proportion of participants
Arm/Group | Intervention Group | Usual Care Group
Number analyzed (Participants) | 7 | 7
proportion of participants | 1 | 1

4. Primary Outcome: The Proportion of Participants That Were Adherent to the Intervention
Description: To determine adherence of a two arm randomized clinical trial of EGCG supplementation in older survivors of cancer by determining the proportion of participants that were adherent to the intervention (taking >70% of study drug).
Time Frame: 12 week
Measure: Number; unit: proportion of participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 7
proportion of participants | 0.857

5. Primary Outcome: Safety of the EGCG Intervention
Description: Total (sum) and severity of adverse events (AEs) reported over 12 weeks of being on study graded using CTCAE v5.0 was determined. Participants were called weekly by study coordinator and asked to report concerns including: symptoms, signs, illnesses, or experiences that develop or worsen during the study. These concerns were graded according to the CTCAE v5.0. Number of participants who reported any AEs during the 12 weeks of the study are reported.
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | Intervention Group | Usual Care Group
Number analyzed (Participants) | 7 | 7
Participants
  Gas/Flatulence-Grade 1 | 2 | 0
  Gas/Flatulence-Grade 2 | 1 | 0
  Constipation-Grade 1 | 1 | 0
  Diarrhea-Grade 1 | 1 | 0
  Indigestion/Dyspepsia-Grade 1 | 1 | 0
  Nausea-Grade 1 | 1 | 0
  Fatigue-Grade 1 | 2 | 2
  Insomnia-Grade 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intervention Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=7) | Usual Care Group (N=7)
Constipation - Grade 1 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea - Grade 1 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Indigestion/Dyspesia - Grade 1 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea - Grade 1 (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue - Grade 1 (General disorders) | 2 (3) | 2 (3)
Insomnia - Grade 1 (Psychiatric disorders) | 2 (4) | 1 (1)
Gas/Flatulence - Grade 1 (Gastrointestinal disorders) | 2 (4) | 0 (0)
Gas/Flatulence - Grade 2 (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT04553666/Prot_SAP_000.pdf